CLINICAL TRIAL: NCT03416231
Title: A Study of Combined Treatment of Apatinib With Docetaxel as Post Second-line Therapy in Advanced Non-squamous Non-small Cell Lung Cancer(NSCLC)
Brief Title: Apatinib Plus Docetaxel in Advanced Non-squamous Non-small Cell Lung Cancer(NSCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Afﬁliated Hospital of North Sichuan Medical College (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APTN-ANSCLC-2017-001
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: NSCLC
Keywords: apatinib; Docetaxel
MeSH Terms: interventions — apatinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib plus docetaxel (Experimental): apatinib combine with docetaxel， 4~6 cycles
  Interventions: Drug: Apatinib; Drug: Docetaxel

INTERVENTIONS:
Drug: Apatinib — apatinib, at a dose of 250 mg daily,Treatment was continued until disease progression.
  Other Names: Aitan
Drug: Docetaxel — Docetaxel, at a dose of 75mg/m2 on days 1 and 22, repeat every 4 weeks for 4~6 cycles.

SUMMARY:
The purpose of this study was to evaluate the effectiveness and safety of apatinib combined with docetaxel in NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female patients, age: ≥ 18 years of age;
* 2. Pathologically diagnosed late (stage IIIB, stage IV, see Annex 1) non-squamous non-small cell lung cancer with measurable lesions (CT scan of tumor lesion longer than 10 mm in diameter, shorter than 15 CT scan of lymph nodes mm, the scanning layer thickness is not more than 5 mm;
* 3. Previous drug treatment consisted of a platinum-based chemotherapy regimen (> 1 chemotherapy regimen) for relapse or failure of treatment.
* 4. The main organs function properly, that is, within 14 days prior to the relevant indicators meet the following requirements:(1) a. Hemoglobin (HB) ≥90 g / L; (no blood transfusion within 14 days):b. neutrophil count (ANC) ≥ 1.5 × 109 / L; c. Platelet count (PLT) ≥80 × 109 / L;(2) biochemical tests to meet the following criteria:a. Total bilirubin (TBIL) <1.5?ULN (upper limit of normal);b. Blood alanine aminotransferase (ALT) and aspartate aminotransferase (AST).

  5. Sign the inform consent form with good compliance.

Exclusion Criteria:

* 1. Squamous cell carcinoma (including adenosquamous carcinoma); Small cell lung carcinoma (including small cell carcinoma and non-small cell mixed lung carcinoma)
* 2. Patients who had previously received docetaxel treatment were excluded
* 3. Patients with active brain metastasis, carcinomatous meningitis, or spinal compression, or disease of brain or pia mater according to the screening test, imaging, CT or MRI tests (patients who have completed the treatment and in a stable condition 21 days before screening could be included, but brain MRI, CT or venography is required to confirm that there are no brain hemorrhage symptoms).
* 4. Patients with uncontrollable hypertension (systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg, despite optimal drug therapy).
* 5. Patients with with grade Ⅱ myocardial ischemia or myocardial infarction, poor control of arrhythmias (including QTc interval male ≥ 450 ms, female ≥470 ms).
* 6. According to NYHA standard, grade Ⅲ ~ Ⅳ heart failure, or cardiac color Doppler ultrasound examination showed left ventricular ejection fraction (LVEF) <50%.
* 7. Coagulation dysfunction (INR> 1.5, PT> ULN +4s or APTT> 1.5 ULN), with bleeding tendency or ongoing thrombolysis or anti-blood coagulation treatment.
* 8. Patients treated with anticoagulation agents or Vitamin K antagonist such as Warfarin, heparin, or other similar drugs.
* 9. Patients who had obvious hemoptysis within 2 months before screening, or experienced daily hemoptysis with a volume more than half a tea spoon (2.5ml) or above.
* 10. Patients who experienced bleeding symptoms of clinical significance within 3 months before screening, or with confirmed bleeding tendency such as hemorrhage of digestive tract, hemorrhagic gastric ulcer, baseline occult blood in stool ++ and above, or vasculitis, etc.
* 11. Patients who manifested arterial/venous thrombus events, e.g. cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism, etc., within 12 months before screening.
* 12. Known genetic or acquired bleeding or bleeding tendency (such as hemophilia, blood coagulation dysfunction, thrombocytopenia, and hypersplenism, etc.).
* 13. Patients who have unhealed wounds or fractures for a long time.
* 14. Patients who received major surgical operations or experienced severe traumatic injuries, bone fracture, or ulcers within 4 weeks before screening.
* 15. Patients with obvious factors affecting absorption of oral drugs, such as difficulties in swallowing, chronic diarrhea and intestinal obstruction, etc.
* 16. Occurrence of abdominal fistula, gastrointestinal perforation, or intraperitoneal abscess within 6 months before screening.
* 17. Patients whose routine urine tests indicate that urine protein ≥ ++ or verifies that the 24-h urine protein quantitation ≥ 1.0 g.
* 18. Patients with active hepatitis B virus or hepatitis c virus infection.
* 19. Active infection requiring antimicrobial treatment, such as antibacterial, antifungal, or antiviral therapy.
* 20. Patients with clinical symptoms, or dropsy of serous cavity requiring surgical treatment (including hydrothorax, ascites, and hydropericardium).
* 21. Patients who have a history of psychotropic drug abuse and are unable to break the habit, or who have a psychogeny.
* 22. Patients who have taken part in other drug clinical tests within 4 weeks before screening.
* 23. Prior VEGFR inhibitor treatment.
* 24. Patients who formerly suffered from or currently are complicated with other uncured malignant tumors, except basal cell carcinoma, carcinoma in situ of cervix and superficial bladder cancer that have been cured.
* 25. Patients who received the treatment with potent CYP3A4 inhibitors within 7 days before screening, or potent CYP3A4 inducers within 12 days before being included.
* 26. Pregnant or lactating women, fertile patients who are unwilling or unable to take effective contraceptive measures.
* 27. Conditions determined by investigators to possibly affect the clinical study or determination of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-11-30 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 6 month
  Proportion of patients with reduction in tumor burden of a predefined amount

SECONDARY OUTCOMES:
progression free survival (PFS) | 12 month
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse.
disease control rate (DCR) | 6 month
  Disease Control Rate (DCR) and Clinical Benefit Rate (CBR) are defined as the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease to a therapeutic intervention in clinical trials of anticancer agents.
6-month overall survival rate | 6 month
  6-month overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Daiyuan Ma, M.D, Principal Investigator — Afﬁliated Hospital of North Sichuan Medical College; xin hu, M.D., Study Director — Nanchong Central Hospital; xiangdong fang, M.d., Study Director — Dazhou Central Hospital
Locations (1):
- Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jiang Q, Zhang NL, Ma DY, Tan BX, Hu X, Fang XD. Efficacy and safety of apatinib plus docetaxel as the second or above line treatment in advanced nonsquamous NSCLC: A multi center prospective study. Medicine (Baltimore). 2019 Jun;98(26):e16065. doi: 10.1097/MD.0000000000016065. PMID 31261514